CLINICAL TRIAL: NCT04078269
Title: Phase I Study of MIDRIXNEO-LUNG, an Autologous Neoantigen-targeted Dendritic Cell Immunotherapy in Patients With Non-small Cell Lung Cancer
Brief Title: MIDRIXNEO-LUNG Dendritic Cell Vaccine in Patients With Non-small Cell Lung Cancer
Acronym: MIDRIXNEO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-04357
Record Dates: First submitted 2019-06-20; First posted 2019-09-06 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: dendritic cell; vaccine; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: intra-patient dose escalation scheme
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC immunotherapy (Experimental): Intra-patient dose escalation of intravenous MIDRIXNEO-LUNG autologous DC vaccine
  Interventions: Biological: Dendritic cell immunotherapy; Biological: Antigen-specific DTH; Biological: Control DTH

INTERVENTIONS:
Biological: Dendritic cell immunotherapy — Intravenous infusions of MIDRIXNEO-LUNG DCs every 2 weeks, using an intra-patient dose escalation scheme progressing along the following range: 10 x10E6 DCs (minimal dose), 20 x 10E6 DCs, 40 x 10E6 DCs, 80 x 10E6 DCs, 100 x 10E6 DCs (maximal dose), until exhaustion of the batch or occurrence of grade ≥3 toxicity event
  Other Names: DC vaccination
Biological: Antigen-specific DTH — Intradermal injection of 1 x 10E6 MIDRIXNEO-LUNG DCs at baseline and after completion of all i.v. DC vaccination rounds. This is used for assessment of induction of antigen-specific immune responses as part of in vivo immunomonitoring (delayed-type hypersensitivity cutaneous reaction as test read-out)
  Other Names: In vivo immunomonitoring - positive test
Biological: Control DTH — Intradermal injection of 1 x 10E6 MIDRIX-CTRL DCs at baseline and after completion of all i.v. DC vaccination rounds. This is used for assessment of background (i.e. non-antigen-specific) reactivity (delayed-type hypersensitivity cutaneous reaction as test read-out)
  Other Names: In vivo immunomonitoring - negative control

SUMMARY:
MIDRIXNEO-LUNG is a novel autologous dendritic cell vaccine for non-small cell lung cancer patients, targeting neoantigens predicted from the patient-individual tumor's mutanome. This first-in-human study aims to primarily establish maximal tolerated dose of MIDRIXNEO-LUNG administered i.v.

DETAILED DESCRIPTION:
Immunotherapy, in the shape of immune checkpoint inhibitors, is now being investigated as an adjuvant therapy in resected NSCLC, with issues unsolved with respect to the optimal duration of treatment, in addition to the unpredictable nature of side-effects with this class of compounds. Also, it is known from advanced disease stages that only a minority of patients respond to checkpoint inhibitors.

An alternative, highly targeted immunotherapeutic approach with an excellent safety track record consists of vaccination. Cancer vaccines aims to prime and/or expand tumor antigen-targeting T-cells and induce immunological memory against later disease relapse. Whereas immune checkpoint blockade boosts inactivated responses of effector T cells, vaccination can potentially activate naive T cells with tumor specificity and in this way broaden the tumor-specific immune responses. However, simple protein-based cancer vaccines have failed in lung cancer so-far, suggesting that the optimal vaccination modality for NSCLC still needs to be established.

Dendritic cells (DCs) are specialized antigen presenting leukocytes that are now recognized as the central controllers of the immune response. The DCs unique capacity to induce robust, highly antigen-specific cytotoxic T-cell responses has led to the use of in vitro-generated autologous DCs as cancer vaccines.

The investigators have developed a novel DC vaccine design that combines robust immunogenicity together with the targeting of patient-tumor specific mutations, also known as neoantigens. The DC vaccine is produced in 2 stages: (1) First, DNA and RNA is isolated from the surgical tumor specimen, sequenced and the sequence is compared to blood cell DNA. In this way, the tumor-specific mutations are identified and the most immunogenic mutated sequences are synthetized. This process takes 3-4 months starting from surgical resection of the tumor. (2) Next, patients undergo a leukapheresis for the harvest of monocytes which are differentiated in vitro into activated DCs. The DCs are finally loaded with the neoantigen-encoding sequences, producing the IMP, MIDRIXNEO.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients older than 18 years with histologically or cytologically proven diagnosis of non-small cell lung cancer, considered functionally operable and surgically resectable (cT1-3 cN0-1 M0 per 8th TNM classification; cT4N0-1 are considered for surgery on a case-by-case basis) and patients considered resectable in an oligometastatic treatment plan
* WHO-ECOG performance status 0 to 2 and absence of any persisting and assessable toxicity > CTC grade 2 due to a previous therapy (surgery and if applicable adjuvant chemotherapy)
* Before patient registration and screening, written informed consent must be given for the interventional study and for the "Prelevation and storage of human tissues and cells" according to ICH/GCP and institutional practice.
* Adequate organ function, including:

  * Adequate bone marrow reserve: absolute neutrophil count > 1.5*10E9/L, platelet count > 100*10E9/L, and Hb > 9.0 g/dL
  * Sufficient renal function as defined by eGFR > 40 ml/min
  * Sufficient hepatic function as defined by total bilirubin ≤1.5× ULN OR direct bilirubin within normal limits for participants with total bilirubin levels >1.5× ULN; AST and ALT ≤ 2.5x ULN
* Having passed all tests defined in the institutional Leukapheresis Donor Fitness Screening, including:

  * Adequate peripheral vein access to perform leukapheresis
  * Adequate coagulation function defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless the participant is receiving anticoagulant therapy
  * Negative test results for HBs-antigen, anti-HBc-serology, anti-HCV serology, anti-HIV1-2 serology, anti-CMV IgM, anti-Syphilis (Treponema pallidum) serology
  * Negative test results for Epstein-Barr virus (IgG and IgM) and for toxoplasmosis (IgG and IgM)
  * For female participants: a negative serum beta-HCG test result less than 1 week before the day of leukapheresis
* For female participants with child-bearing potential, the willingness to follow contraceptive guidance and pregnancy testing during the projected duration of the trial (see Appendix B on Contraceptive Guidance and Pregnancy Testing)
* For male participants having a partner with child-bearing potential: agreement to use contraception during the projected duration of the trial, starting with the screening visit through 90 days after the last dose of trial treatment. Sperm donation must have been performed before anti-cancer treatment as per standard practice

Exclusion Criteria:

* Presence of oncogenic driver genomic alterations for which a targeted therapy is available
* Concomitant participation in another clinical interventional trial
* Prior treatment with autologous or allogeneic dendritic cell-based vaccines
* Prior malignancy, except for adequately treated basal cell, superficial or in situ cancer of the bladder or the cervix, or other cancer for which the patient has been disease-free for at least five years.
* Dermatological pathology interfering with the in vivo immunomonitoring readout (DTH skin test)
* Disease requiring chronic treatment with systemic glucocorticosteroids with a daily dose > 10 mg oral prednisolone or equivalent, or other immunosuppressive drugs. Inhaled corticosteroids and topical corticosteroids on skin sites other than those used for DTH are allowed.
* Chronic or active concomitant infection requiring active therapy, including including HIV, viral hepatitis (HBV, HCV), CMV or fungal infection
* Autoimmune disease requiring active treatment at the time of the study
* Organ allograft
* Chronic comorbidity (such as asthma, COPD, heart failure, renal failure, arterial hypertension or diabetes mellitus) that is uncontrolled or not stabilized under medication at the time of study enrollment, OR stable yet severe enough to constitute an unwarranted high risk for the investigational cellular therapy.
* For female participants: pregnancy or lactation, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 90 days after the last dose of trial treatment
* Any organic brain syndrome or other significant psychiatric abnormality which would comprise the ability to give informed consent and preclude participation in the full protocol and follow-up.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of preparing and administrating the autologous dendritic cell-based vaccine in surgically-treated non-small cell lung cancer patients | From the day of leukapheresis until 3-4 weeks after the last vaccine dose level, i.e. 3 to 5 months depending on the number of doses that can be administered
  Toxicity measures as defined by common toxicity criteria v5.0. The maximal tolerated and/or feasible dose will be defined from the intra-patient dose excalation scheme

SECONDARY OUTCOMES:
Feasibility of producing sufficient dendritic cell for vaccination in surgically treated NSCLC | From the day of enrollment prior to surgery until the last vaccine dose level, i.e. 2 to 4 months depending on the number of doses that can be administered
  Success rate (%) of producing sufficient dendritic cells for vaccination
Biological activity of the vaccine (elicitation of immune responses against vaccine neoantigens) in vitro | From the day of leukapheresis until 3-4 weeks after the last vaccine dose level, i.e. 3 to 5 months depending on the number of doses that can be administered. Whenever possible, repeat testing will be performed 3 and 6 months after vaccination.
  Vaccine-induced immunological responses as measured by in vitro immunomonitoring assays
Biological activity of the vaccine (elicitation of immune responses against vaccine neoantigens) in vivo | From the day of leukapheresis until 3-4 weeks after the last vaccine dose level, i.e. 3 to 5 months depending on the number of doses that can be administered. Whenever possible, repeat testing will be performed 3 and 6 months after vaccination.
  Vaccine-induced immunological responses as measured by in vivo immunomonitoring test (delayed-type hypersensitivity skin reaction)
Clinical activity of this type of vaccine as reflected by relapse-free survival (months) | From the day of leukapheresis onwards during 2 years
  Relapse-free survival based on clinical and/or radiological event

CONTACTS AND LOCATIONS:
Overall Officials: Karim Y Vermaelen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brabants E, Heyns K, De Smet S, Devreker P, Ingels J, De Cabooter N, Debacker V, Dullaers M, VAN Meerbeeck JP, Vandekerckhove B, Vermaelen KY. An accelerated, clinical-grade protocol to generate high yields of type 1-polarizing messenger RNA-loaded dendritic cells for cancer vaccination. Cytotherapy. 2018 Sep;20(9):1164-1181. doi: 10.1016/j.jcyt.2018.06.006. Epub 2018 Aug 16. PMID 30122654